CLINICAL TRIAL: NCT03472183
Title: Exploration of the Enteric Nervous System in Alzheimer Disease : a Monocentric Pilot Study
Brief Title: Exploration of the Enteric Nervous System in Alzheimer Disease
Acronym: SYNEMA
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no patients included
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RC17_0252
Record Dates: First submitted 2018-02-28; First posted 2018-03-21 (Actual); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Alzheimer Disease
Keywords: Enteric nervous system; Alzheimer disease; biomarker; colonic biopsies; neurodegenerative disease
MeSH Terms: conditions — Alzheimer Disease; Neurodegenerative Diseases

STUDY DESIGN:
Intervention Model Description: 3 types of patients will be included:
  * 10 patients with Alzheimer's disease and as controls:
  * 10 patients with Parkinson's disease
  * 10 patients without neurodegenerative disease.
  During the course of the colonoscopy that these 30 patients should have in the context of their medical usual care, additionnal biopsies of colon will be removed to perform in vitro analysis for this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients with Alzheimer's disease (Other): During the course of the colonoscopy that the patients should have in the context of their usual medical care, additional biopsies of colon will be removed to perform in vitro analysis for this study.
  Interventions: Other: biopsies of colon
- Patients with Parkinson's disease (Other): During the course of the colonoscopy that the patients should have in the context of their usual medical care, additional biopsies of colon will be removed to perform in vitro analysis for this study.
  Interventions: Other: biopsies of colon
- Patients without neurodegenerative disease (Other): During the course of the colonoscopy that the patients should have in the context of their usual medical care, additional biopsies of colon will be removed to perform in vitro analysis for this study.
  Interventions: Other: biopsies of colon

INTERVENTIONS:
Other: biopsies of colon — Removal of additional biopsies of colon during the course of a colonoscopy planned for usual medical follow-up of patient

SUMMARY:
The close homology between the central and enteric nervous system suggests that a disease process affecting the central nervous system could also involve its enteric counterpart. This has already been demonstrated for patients with Parkinson's disease but needs to be proven for Alzheimer's disease. Studies on enteric nervous system during Alzheimer's disease are indeed in low number and don't have led to definite conclusion. The investigators thus propose to realize a complete analysis of the enteric nervous systems in Alzheimer's disease by studying the presence of "tau' protein, of beta-amyloid peptide,...

not only by immunohistochemical but also by a biochemical approach. This study will be realized from colonic samples.

DETAILED DESCRIPTION:
The close homology between the central and enteric nervous system suggests that a disease process affecting the central nervous system could also involve its enteric counterpart. The investigators have recently shown in that the enteric neurons can be readily analyzed using routine colonic biopsies. The investigators propose that the enteric nervous system could represent a unique window to assess the neuropathology in living patients with a neurodegenerative disorder. The investigators have already used this approach to show that Parkinson's disease pathology was recapitulated in a single colonic biopsy. By contrast to Parkinson's disease, the detection of Alzheimer's disease pathology in the enteric neurons has so far failed. This may be due to the low number of human tissue samples in addition to the low sensitivity of the immunohistochemical methods that were used. The aim of the current research project will be therefore to reevaluate Alzheimer's disease pathology in a large number of human colonic samples using both a morphological and biochemical approach.

The Hypothesis is that the enteric nervous system could represent a unique window to assess the neuropathology in living patients with Alzheimer's disease. This might open the way to the development of novel Alzheimer's disease biomarkers that will directly assess the neuropathological process.

ELIGIBILITY:
Inclusion Criteria:

* For the 3 groups of patients : colonoscopy planned by a gastroenterologist in the context ot the usual medical follow-up of the patient

For patients with Alzheimer's disease :

* Patient with early to moderate Alzheimer disease (continuum of patients with mild cognitive impairment due to Alzheimer's disease and patients diagnosed with probable Alzheimer's disease) according to the National Institute of Aging-Alzheimer's Association (NIA AA) criteria
* Mini-Mental State Examination (MMSE) score ≥18;
* Has one informant or care partner;
* No parkinsonian syndrome
* No sign of lewy Body dementia

For patients with Parkinson's disease:

* patients with Parkinson Disease according to the United Kingdom Parkinson's Disease Society Brain Bank (UKPDSBB) criteria
* No dementia sign or cognitive deficit associated to Alzheimer's disease

For patients without neurodegenerative disease:

* No history or current neurological/degenerative condition (e.g, lewy body dementia, Parkinson's disease, Parkinsonian syndrome, Alzheimer's disease,…)
* No memory complaint with a Mac Nair score ≤15
* MMSE score ≥28 ;
* Patient at risk of colic cancer with a colonoscopy scheduled

Exclusion Criteria:

For the 3 groups of patients : :

* History of colonic disorder ((e.g inflammatory condition, adenocarcinoma)
* contra-indications to colonoscopy

For patients with Alzheimer's disease and for patients with Parkinson's disease:

- Any neurological/neurodegenerative condition different from the group to which it belongs (e.g other than Alzheimer's disease for Alzheimer's disease group or other than Parkinson's disease for Parkinson's disease group….)

For patients without neurodegenerative disease:

* Any neurological/neurodegenerative condition (e.g lewy body dementia, Parkinsonian syndrome, Parkinson's disease, Alzheimer's disease..)..
* functional colopathy

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-04-26 (Actual); Primary Completion 2019-09-18 (Actual); Study Completion 2019-09-18 (Actual)

PRIMARY OUTCOMES:
Differences in extracellular deposits of beta-amyloid peptide in the enteric nervous system between patients with Alzheimer's disease, patients with Parkinson's disease and patients without neurodegenerative disease. | colonoscopy performed within 3 months after inclusion in the study
  In vitro analysis of the presence of beta-amyloid peptide in biopsies of colon from patients with Alzheimer's disease ans as controls from patients with Parkinson's disease and from patients without neurodegenerative disease

SECONDARY OUTCOMES:
Differences in tau protein in the enteric nervous system between patients with Alzheimer's disease, patients with Parkinson's disease and patients without neurodegenerative disease. | within 3 months after inclusion
  In vitro analysis of the presence of tau protein in biopsies of colon from patients with Alzheimer's disease ans as controls from patients with Parkinson's disease and from patients without neurodegenerative disease
Differences in neuronal loss in enteric submucosal tissue between patients with Alzheimer's disease, patients with Parkinson's disease and patients without neurodegenerative disease | within 3 months after inclusion
  In vitro analysis of the presence of neuronal loss in biopsies of colon from patients with Alzheimer's disease ans as controls from patients with Parkinson's disease and from patients without neurodegenerative disease
Differences in neuronal Glia cells in the enteric nervous system between patients with Alzheimer's disease, patients with Parkinson's disease and patients without neurodegenerative disease. | within 3 months after inclusion
  In vitro analysis of the presence neuronal glia cells in biopsies of colon from patients with Alzheimer's disease ans as controls from patients with Parkinson's disease and from patients without neurodegenerative disease

CONTACTS AND LOCATIONS:
Overall Officials: Pascal DERKINDEREN, Pr, Principal Investigator — Nantes University Hospital